CLINICAL TRIAL: NCT06938412
Title: Exercise Activity Intervention With Sensor-Based Engagement in Patients With Atrial Fibrillation (EASE-AF)
Brief Title: Exercise Activity Intervention With Sensor-Based Engagement in Patients With Atrial Fibrillation
Acronym: EASE-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Janice.Chyou, Assistant Clinical Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-00464; 24SCEFIA1249819 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases
Keywords: Atrial Fibrillation; Physical Activity; Exercise; Digital Health Intervention; Wearable Technology; Symptoms; Quality of Life
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients With Atrial Fibrillation (Experimental): Patients with symptomatic, paroxysmal AF.
  Interventions: Device: Physical Activity Intervention Using FitBit Wearable Device

INTERVENTIONS:
Device: Physical Activity Intervention Using FitBit Wearable Device — The intervention is a digital technology-driven, patient-centric approach to physical activity and exercise intervention with tailored digital engagement and progressive physical activity goals (the intervention). The intervention will be conducted using FitBit wearable device.

SUMMARY:
Atrial fibrillation (AF) affects 1 in 4 individuals during their lifetime and continues to increase in frequency and impact. Exercise intervention has established benefits to improve AF symptoms and burden in clinical studies. However, lack of access to exercise programs has limited therapeutic adoption. The growth of technology-driven health care and diagnostics, recognized as an emerging priority by the American Heart Association, offers an opportunity for a pragmatic and patient-centered approach to meet this need. EASE-AF is a prospective, interventional study with a sequential run-in control to evaluate if a digital health-driven, patient-centered exercise intervention improves AF symptoms and burden. The research team will enroll 120 patients with symptomatic, paroxysmal AF. The main impact of this study will be the establishment of evidence for a novel, pragmatic paradigm for a patient-centered, digital technology-driven personalized exercise intervention for patients with AF.

ELIGIBILITY:
Inclusion Criteria:

* ≥40years of age
* Paroxysmal AF
* Electrocardiographic (or equivalent) documentation of AF within 12 months (would need to have evidence of AF after initial post-ablation blanking period if the patient had prior AF ablation)
* AF Severity Scale (AFSS) symptom score 13-26
* Self-report weekly moderate-vigorous physical activity (MVPA) 30-120 minutes

Exclusion Criteria:

* Unable to give consent
* ≤90 days from AF ablation, coronary revascularization, heart failure hospitalization
* Left ventricular ejection fraction (LVEF) <50%, moderate to severe stenotic valvular heart disease or severe regurgitant valvular disease or history of mechanical valve replacement, presence of implanted pacemaker or defibrillator system
* Labile INR or unable to take anticoagulant despite indication
* Life expectancy < 1 year
* Hemodialysis; severe pulmonary or liver disease
* Musculoskeletal, balance/gait issues, severe peripheral vascular disease, or neuropathy or other neurologic conditions limiting exercise
* Self-report MVPA <30 minutes
* Upon initial screening, if the participant's baseline FitBit-measured MVPA ≥180 minutes/week (despite self-report range of 30-120 minutes), the participant will be further excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation Severity Scale (AFSS), Symptom Severity Domain | Baseline, End of 4-week Run-in Control Period, End of 24-week Physical Activity Intervention Period
  The Symptom Severity domain (Part C) of the validated Atrial Fibrillation Severity Scale (AFSS) questions patients regarding the severity of 7 AF-related symptoms (on scale of 0-5 per question, 5 denoting a great deal of symptom and 0 with no symptom) over the preceding 4-week period. Total scores range 0-35 on the Symptom Severity Domain of the Atrial Fibrillation Severity Scale (AFSS), higher score denotes more severe AF-related symptoms.

SECONDARY OUTCOMES:
Atrial Fibrillation Severity Scale (AFSS) | Baseline, End of 4-week Run-in Control Period, End of 24-week Physical Activity Intervention Period
  The full Atrial Fibrillation Severity Scale (AFSS) is composed of 19-items, investigating four domains: global well-being, symptom burden, health care utilization, symptom severity.
  Global well-being: 1-10; 10 denotes best possible quality of life. Symptom burden: Composite of AF burden as AF duration + AF frequency + AF severity; ranging 0-30, higher denotes more symptom burden.
  Health care utilization: ER visits (0-7, higher number denotes more utilization), Hospitalizations (0-7, higher number denotes more utilization), Specialist visits (0-7, higher number denotes more utilization); Symptom Severity: 0-35, higher score denotes more severe AF-related symptoms
AF Arrhythmia Burden: Percentage of time in AF | Baseline, End of 4-week Run-in Control Period, End of 24-week Physical Activity Intervention Period
  Global AF arrhythmia burden will be measured as percentage of time in AF measured during an 8-14-day monitoring period at the end of each time point as quantified by either clinically validated patch-based monitoring system or loop recorder.
AF Arrhythmia Burden: Duration of longest AF Arrhythmia Episode | Baseline, End of 4-week Run-in Control Period, End of 24-week Physical Activity Intervention Period
  Duration of the longest AF episode during the monitoring period will be quantified by either clinically validated patch-based monitoring system or loop recorder.
Weekly Step Counts | Baseline, End of 4-week Run-in Control Period, End of 24-week Physical Activity Intervention Period
  Weekly step counts measured by FitBit wearable device provided by the study
Weekly Exercise Minutes | Baseline, End of 4-week Run-in Control Period, End of 24-week Physical Activity Intervention Period
  Weekly exercise minutes measured by FitBit wearable device provided by the study

CONTACTS AND LOCATIONS:
Overall Officials: Janice Y Chyou, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Not planning to share individual participant data. Aggregate data will be shared instead.